CLINICAL TRIAL: NCT02711462
Title: A Phase 1, Double Blind, Third-Party Open, Randomized, Placebo Controlled, Single And Multiple Dose, Parallel Group Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PF-06687234 In Healthy Subjects
Brief Title: Study in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-06687234
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was prematurely terminated on 06 October 2016 due to the potential risk of further dosing in healthy subjects
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B7581001; 2015-000710-22 (EudraCT Number); DEKAVIL (Other: Alias Study Number)
Record Dates: First submitted 2016-01-08; First posted 2016-03-17 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Cohort 1 (Other): Subjects will receive 2mg of PF 06687234 or placebo via the SC route
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 2 (Other): Subjects will receive 20mg PF 06687234 or placebo via the SC route
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 3 (Other): This is an optional cohort that may be added anytime during the study. In this cohort, subjects will receive PF 06687234 or placebo via the SC route
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 4 (Other): Subjects will receive 40mg of PF 06687234 or placebo via the SC route
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 5 (Other): Subjects will receive 80mg of PF 06687234 or placebo via the SC route
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 6 (Other): Subjects receive a single dose of PF 06687234 or placebo via the IV route
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 7 (Other): This is an optional cohort where Japanese subjects will receive PF 06687234 or placebo via the SC route
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 8 (Other): Subjects in this cohort may receive 20 mg of PF 06687234 or placebo via the SC route every week with a total of 5 doses
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 9 (Other): Subjects in this cohort may receive 40 mg of PF 06687234 or placebo via the SC route every two weeks with a total of 3 doses
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 10 (Other): This is an optional cohort. The maximum dose tested in the multiple dose cohort will not exceed the highest dose tested in the single dose cohorts
  Interventions: Drug: PF-06687234; Drug: Placebo
- Cohort 11 (Other): This is an optional cohort. The maximum dose tested in the multiple dose cohort will not exceed the highest dose tested in the single dose cohorts
  Interventions: Drug: PF-06687234; Drug: Placebo

INTERVENTIONS:
Drug: PF-06687234 — PF-06687234 will be administered via the SC or the IV route and in either single dose or multiple doses
  Other Names: Dekavil
Drug: Placebo — In Cohorts 1 and 2, up to 1 subject will receive placebo. In all other Cohorts (Cohorts 3 to 11), up to 2 subjects will receive placebo.

SUMMARY:
This Phase 1 study will be a double blind, third party open (ie, subject blind, investigator blind and Sponsor open), randomized, placebo controlled, single and multiple dose escalation study in healthy subjects, females of non childbearing potential and males between the ages of 18 and 55 years, inclusive. There may be up to 11 Cohorts in the study. Approximately 7 cohorts are anticipated in the Single Dose (SD) portion of the study and up to 4 cohorts are anticipated in the Multiple Dose (MD) portion of the study.

Following the last subject Day 28 visit from the first two single dose cohorts (Cohorts 1 and 2), all available data inclusive of Day 28 will be evaluated for PK, immunogenicity, safety and tolerability. FDA review and agreement to move forward will take place before the remaining single dose cohorts and the multiple dose phase (Cohorts 3 to 11) can be initiated.

A total of up to approximately 82 subjects are anticipated to be enrolled in the study. The duration of dosing in the multiple dose cohorts would be 4 weeks and the regimen may include weekly (total of 5 doses), every 2 weeks (total of 3 doses) or monthly dosing (total of two doses).

ELIGIBILITY:
INCLUSION CRITERIA

* Healthy females of non childbearing potential and healthy males
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)
* Ability to personally sign and date the informed consent document and able to comply with schedule of activities
* For Single Dose Cohort 7 only, Japanese subjects must have four biological Japanese grandparents born in Japan.

EXCLUSION CRITERIA

* Evidence or history of clinically significant health concerns
* Treatment with an investigational drug within 30 days
* Exposure to any live vaccines within 28 days prior to investigational product administration.
* History of drug and/ or alcohol abuse and tobacco use equivalent of 5 cigarettes per day.
* Known history of infection with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus
* Pregnant female subjects
* History of sensitivity to heparin
* Unwilling or unable to comply with the Lifestyle Guidelines as stated in the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | 4 weeks in the single dose portion and 8 weeks in the multiple dose portion
  To determine the safety and tolerability of PF 06687234 by assessing averse events, vital signs measurements, 12 lead ECGs, physical examination findings, blood and urine safety tests including ferritin, transferrin, serum iron, reticulocytes, hemoglobin, platelets and any abnormal laboratory results.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF 06687234 (IV and SC single doses) | Day 1 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose and 8 and 11 days post dose along with early termination or follow up visit.
Maximum Observed Plasma Concentration (Cmax) of PF 06687234 (SC multiple doses) | Day 1 and Day 29 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose. Pre-dose samples on Day 8, 15, 22, 36, 39 and 43 along with early termination or follow up visit.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF 06687234 (IV and SC single doses) | Day 1 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose and 8 and 11 days post dose along with early termination or follow up visit.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF 06687234 (SC multiple doses) | Day 1 and Day 29 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose. Pre-dose samples on Day 8, 15, 22, 36, 39 and 43 along with early termination or follow up visit.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF 06687234 (IV and SC single doses) | Day 1 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose and 8 and 11 days post dose along with early termination or follow up visit.
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF 06687234 (SC multiple doses) | Day 1 and Day 29 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose. Pre-dose samples on Day 8, 15, 22, 36, 39 and 43 along with early termination or follow up visit.
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF 06687234 (IV and SC single doses) | Day 1 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose and 8 and 11 days post dose along with early termination or follow up visit.
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF 06687234 (SC multiple doses) | Day 1 and Day 29 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose. Pre-dose samples on Day 8, 15, 22, 36, 39 and 43 along with early termination or follow up visit.
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast
Plasma Decay Half-Life (t1/2) of PF 06687234 (IV and SC single doses) | Day 1 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose and 8 and 11 days post dose along with early termination or follow up visit.
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Plasma Decay Half-Life (t1/2) of PF 06687234 (SC multiple doses) | Day 1 and Day 29 prior to 0 hr & 0.5, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96 hours post dose. Pre-dose samples on Day 8, 15, 22, 36, 39 and 43 along with early termination or follow up visit.
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Incidence of development of anti-drug antibody (ADA) | up to 2 months
Incidence of development of neutralizing antibody (NAb) | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Laure Mendes da Costa, Principal Investigator — Pfizer Clinical Research Unit
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7581001&StudyName=A%20Phase%201%2C%20Double%20Blind%2C%20Third-party%20Open%2C%20Randomized%2C%20Placebo%20Controlled%2C%20Single%20And%20Multiple%20Dose%2C%20Parallel%20Group%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20And%20Pharmacodynamics%20Of%20Pf-06687234%20In%20Healthy%20Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7581001&StudyName=A+Phase+1%2C+Double+Blind%2C+Third-party+Open%2C+Randomized%2C+Placebo+Controlled%2C+Single+And+Multiple+Dose%2C+Parallel+Group+Study+To+Evaluate+The+Safety%2C+Tolerability%2C+Pharmacokinetics%2C+And+Pharmacodynamics+Of+Pf-06687234+In+Healthy+Subjects